CLINICAL TRIAL: NCT06316037
Title: Adaptation of Work in a Hospital Environment and Assessment of Feelings of Quality of Life at Work, Teleworking and Face-to-face
Brief Title: Adaptation of Work in a Hospital and Assessment of Feelings of Quality of Life at Work, Teleworking and Face-to-face
Acronym: ADAPTAWORK_2
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2024 DUTHEIL ADAPTAWORK_2
Record Dates: First submitted 2024-03-06; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Work-Related Stress; Work-Related Condition
Keywords: Teleworking; working at home
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ADAPTAWORK_2 study is a follow-up to the first qualitative study, to evaluate the feelings of hospital workers in all occupations about teleworking. This involves measuring the variation between three periods: before the COVID-19 pandemic, during the first lockdown an after the pandemic.

Secondary objectives were: 1) to evaluate wich factors were associated to the feelings towards teleworking, 2) to assess musculo-squeletal disorders among teleworkers and the other participants, 3) to assess psycho-social risks among teleworkers and the oher participants, and 4) to evaluate teleworking costs

DETAILED DESCRIPTION:
This is a quantitative study carried out at the Clermont-Ferrand University Hospital and in the Hospital Centers of the Homogenous Territorial Group (HTG). The target population was made up of all hospital workers in these establishments who agreed to participate and complete the online questionnaire, regardless of their function or grade in the work establishment.

ELIGIBILITY:
Inclusion Criteria:

* all hospital workers in the University Hospital Centre of Clermont-Ferrand, and the hospitals belonging to the same HTG who agreed to participate and complete the questionnaire, regardless of their function or grade in the work establishment

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital workers
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Feeling about teleworking | Period 1 of questionnaire= from March 17, 2019 to March 17, 2020; Period 2=from March 18, 2020 to January 18, 2021; Period 3= from January 19, 2021 to January 20, 2024 (study end date).
  visual analogic scale (VAS), from 0 (very bad feeling) to 100 (very good feeling) scale

SECONDARY OUTCOMES:
Musculo-squeletic pain | Period 3= from January 19, 2021 to January 20, 2024 (study end date).
  Using the NORDIC questionnaire, participants could express their pain in person or by teleworking
psychosocial risks | Period 3= from January 19, 2021 to January 20, 2024 (study end date).
  VAS scales from 0 to 100
purchases | Period 1 of questionnaire= from March 17, 2019 to March 17, 2020; Period 2=from March 18, 2020 to January 18, 2021; Period 3= from January 19, 2021 to January 20, 2024 (study end date).
  self questionnaire about the purchases they have made in order to telework, and the approximate cost of these purchases

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No
It was not planned to share participants' IDs, which only the investigator is able to know.